CLINICAL TRIAL: NCT07003334
Title: Correlation of Psychological Distress With Efficacy of Immune Checkpoint Inhibitors in Patients With Advanced Gastric Cancer
Brief Title: Correlation of Psychological Distress and Immune Checkpoint Inhibitors in Gastric Cancer
Acronym: PDICI
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-362; Nanfang Hospital (Registry Identifier: Nanfang Hospital)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancers
Keywords: Psychological Distress; Immune Checkpoint Inhibitors; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum cortisol， Adrenocorticotropic Hormone (ACTH)，Plasma epinephrine (Epi)，Norepinephrine (NE)，Serotonin (5-HT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric cancer patients who plan to reveive immune checkpoint inhibitors treatment: As this was an observational study, no additional visits or laboratory analyses or assessments other than those required by routine, clinical practice were required. Patients must sign an updated informed consent form (ICF- approved by Ethics Committeettee) before performing data collection. After obtaining the patient's informed consent, the patient's clinical routine diagnosis and treatment information will be collected; We collected psychological assessment questionnaires, quality of life assessment questionnaires, serum cortisol, corticotropin (ACTH) , plasma epinephrine (Epi) , and noradrenaline (NE) 、serotonin along with clinical diagnosis and treatment nodes, data, the number and time of the study visits were according to the time points of the routine clinical patient review ( peritoneal exploration for advanced gastric cancer, 4 cycles of immunotherapy/combined chemotherapy before surgery, surgery, treatments after surgery) .

SUMMARY:
1. Background Gastric cancer (GC) is a leading global cause of cancer-related mortality, with over 1 million new cases and 769,000 deaths in 2020. In China, 80% of patients present with advanced disease, for whom perioperative chemotherapy, surgery, and lymphadenectomy are standard. Recent phase III trials (Checkmate-649, KEYNOTE-062, ORIENT-16) demonstrate that immune checkpoint inhibitors (ICIs) combined with chemotherapy improve progression-free survival (PFS: 2.8-10.5 months) and overall survival (OS: 11.1-18.4 months) compared to chemotherapy alone. However, outcomes remain suboptimal, necessitating exploration of novel predictive biomarkers and resistance mechanisms.

   Emerging evidence implicates chronic stress in cancer progression and treatment response. Chronic stress activates the hypothalamic-pituitary-adrenal (HPA) axis and sympathetic nervous system, elevating cortisol, catecholamines, and glucocorticoids. These hormones suppress immune function by reducing CD8+ T cells and natural killer (NK) cell activity while increasing immunosuppressive cells (e.g., regulatory T cells, myeloid-derived suppressor cells). Preclinical studies link chronic stress to metastasis via extracellular trap (NET) formation, impaired antitumor immunity, and resistance to PD-1/PD-L1 blockade. Clinically, chronic stress correlates with worse survival in non-small-cell lung cancer patients receiving ICIs. Despite these findings, psychological screening remains underutilized in oncology. This study aims to investigate the impact of chronic stress on ICI efficacy in advanced gastric cancer.
2. Objectives

   Primary Objective:

   Evaluate the association between chronic stress and tumor response (via Tumor Regression Grade, TRG) in advanced gastric cancer patients undergoing neoadjuvant immunotherapy.

   Secondary Objectives:

   Assess the effect of chronic stress on post-gastrectomy quality of life (QoL).

   Analyze correlations between chronic stress biomarkers and survival outcomes (PFS, OS).
3. Study Endpoints

   Primary Endpoint:

   Pathological response assessed by TRG (Mandard criteria).

   Secondary Endpoints:

   QoL (EORTC QLQ-C30/STO22 questionnaires).

   PFS and OS.

   Exploratory Endpoints:

   Dynamic changes in chronic stress biomarkers (serum cortisol, ACTH, epinephrine, norepinephrine, serotonin).

   Correlation of biomarker levels with TRG and survival.
4. Study Design Type: Single-center, prospective observational study. Duration: 36 months. Sample Size: 268 patients (134 high chronic stress, 134 low chronic stress).

   Inclusion Criteria:

   Age 18-75 years.

   Histologically confirmed gastric adenocarcinoma (per Japanese Gastric Cancer Guidelines, 2017).

   Scheduled for neoadjuvant immunotherapy + radical gastrectomy.

   Informed consent.

   Exclusion Criteria:

   Pregnancy/breastfeeding.

   Prior upper abdominal surgery (excluding cholecystectomy).

   Active infection, autoimmune disease, or corticosteroid use within 1 month.

   Psychiatric disorders or investigator-deemed unsuitability.

   Withdrawal Criteria:

   Patient request, loss to follow-up, or safety concerns.
5. Methods

   Chronic Stress Assessment:

   Validated psychological questionnaires (e.g., Hospital Anxiety and Depression Scale) at baseline and treatment milestones.

   Biomarker analysis: Serum cortisol, ACTH, epinephrine, norepinephrine, serotonin at key timepoints (pre-treatment, post-neoadjuvant therapy, post-surgery).

   Clinical Data Collection:

   TRG evaluation post-surgery.

   QoL assessments at 1, 3, 6, 12, 18, 24, and 36 months post-surgery.

   Survival tracking via hospital records and follow-up visits.

   Statistical Analysis:

   Stratification by baseline stress scores (high/low).

   Cox regression for survival outcomes; logistic regression for TRG-QoL correlations.

   Significance threshold: *p* < 0.05.
6. Significance This study addresses a critical gap in understanding how psychological factors modulate ICI efficacy. By identifying chronic stress as a predictor of treatment response, results may guide personalized interventions (e.g., beta-blockers, behavioral therapy) to improve outcomes in advanced gastric cancer.

DETAILED DESCRIPTION:
Gastric carcinoma (GC) remains a globally important cancer, with more than one million new cases and an estimated 769,000 deaths in 2020(equivalent to one in every 13 deaths worldwide) , it ranks fifth globally in incidence and fourth globally in mortality [1] . In China, 80% of gastric cancer patients are advanced, and the standard recommendation for locally advanced gastric cancer is perioperative adjuvant chemotherapy plus standard gastrectomy plus radical lymphadenectomy [2,3] . A series of large phase III studies (including Checkmate-649, ATTRACTION-04, KEYNOTE-062, ORIENT-16[4,5,6,7]) of completed ICI plus chemotherapy in gastric/esophageal/GEJ cancer showed a median PFS of 2.8 to 10.5 months for patients treated with ICI plus chemotherapy, median OS was 11.1-18.4 months. For advanced gastric/oesophagogastric junction gastric/oesophagogastric cancer, immunotherapy combined with chemotherapy versus first-line chemotherapy resulted in clinically meaningful PFS benefit, improved and durable objective responses, maintenance of HRQOL, and improved survival, also acceptable safety profile [4,5,6,7] , but the prognosis of advanced gastric cancer remains poor. There is still a lot of room for exploration to improve the efficacy of adjuvant therapy. It is imperative to find new predictive markers of immunotherapy efficacy, and explore the mechanism of drug resistance to immune checkpoint inhibitors.

In addition to genetic and tumor microenvironmental factors, psychological factors may also play a role in cancer treatment [8] . Chronic stress refers to the persistent non-specific adaptive response of the body triggered by the activation of the hypothalamic-pituitary-adrenal, glandular axis and sympathetic nervous system under the stimulation of physiological and psychological stressors, anxiety and depression. Chronic stress can affect the functioning of the immune system [9,12,13] . Related studies have shown that there may be different mechanisms by which chronic stress affects the progression and treatment of gastric cancer: depression induces neuroendocrine phenotypes through the catecholamine/β2-AR/MACC1 axis, thereby accelerating the invasion and metastasis of gastric cancer [6] ; Chronic stress, which activates the hypothalamic-pituitary-adrenal axis as well as the sympathetic nervous system, causes increased levels of cortisol, adrenergic hormones, the glucocorticoid released during chronic stress leads to the formation of NETs (extracellular traps) and the establishment of a microenvironment that promotes metastasis, which may contribute to the development of metastatic lesions, whereas digestion of NETs with DNase I in experimental mice prevents chronic stress-induced metastasis [11] . The stress-glucocorticoid-tsc22D3 axis can impair therapy-induced, antitumor immunity [12] . Preclinical studies have shown that pain-induced activation of the HPA axis and subsequent glucocorticoid, release can elicit anti-inflammatory effects, including apoptosis of T lymphocytes and neutrophil [13] . Endogenous glucocorticoids, the persistent release of hormones, also inhibit antigen presentation, further undermining systemic immune function [13] . In a large number of animals, studies have shown that exposure to chronic stress causes depression-like and anxiety-like symptoms in mice, thereby promoting tumor progression and metastasis [14,15,16] . Stress hormones can directly affect the malignant molecular characteristics of tumor cells [14,17,18] . Preclinical studies have shown that chronic stress also plays a potential role in promoting the development of the immunosuppressive tumor microenvironment [14,19,20] . Chronic stress exposure reduces CD8 + T cells and natural killer cells Proportion of cells and inhibit their function, while also increasing the infiltration of immunosuppressive cells such as regulatory T cells and myeloid-derived suppressor cells [12,19,21] . In mouse tumor models, studies have shown that chronic stress impairs the response to programmed cell death-1(PD-1)/PD-L1 blockade [12,22] . Chronic stress is also strongly associated with cancer, patient outcomes, and survival outcomes, as those with symptoms of depression or anxiety are at increased risk of relapse and Mortality[23]. However, screening and monitoring of psychological status in the clinic is often neglected and is not part of the current diagnosis and treatment routine [14] .

As immunotherapy becomes the cornerstone of treatment, it is crucial and important to study the relationship between chronic stress and the efficacy of ICIs. Studies have shown an association between chronic stress and worse clinical prognosis in patients with advanced non-small-cell lung carcinoma treated with ICIS, which highlights the potential significance of chronic stress in cancer management [24] . A 2020 study found that in colorectal cancer, β receptor and COX2 inhibition by preoperative propranolol/Idolac improved tumor metastasis, immunity, and inflammatory response-related markers [25] ; Similar results have been reported in breast cancer [26,27] . Psychological distress may have some predictive power for selected cancer presentations, including gastric cancer [28] . However, for gastric cancer, clinical evidence supporting the relationship between chronic stress and ICIS efficacy is limited, underscoring the need for prospective clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent;
* 18≦ age ≦75 years;
* Sex: no limitation;
* Patients with gastric adenocarcinoma diagnosed according to the 15th edition of the Japanese gastric cancer statute, 2017, after endoscopic biopsy of the primary lesion;
* Patients requiring preoperative immune checkpoint inhibitor therapy at the discretion of the treating physician, followed by radical gastrectomy.

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Serious mental illness;
* History of upper abdominal surgery (except for laparoscopic cholecystectomy) ;
* Patients with gastric cancer who do not wish to undergo neoadjuvant immunotherapy;
* Patients with a history of continuous systemic corticosteroid therapy within the past 1 month;
* Patients with active infection, active or refractory autoimmune disease, or uncontrolled systemic disease;
* Patients at the discretion of the investigator, were deemed unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was patients with gastric cancer who were scheduled for laparoscopic gastrectomy after preoperative immunotherapy.
Sampling Method: Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Regression Grade （TRG） | 7 Days
  Tumor Regression Grade (TRG) is a histopathological scoring system used to assess the degree of tumor response to neoadjuvant therapy (e.g., chemotherapy or radiation) in resected specimens. It quantifies residual viable tumor cells versus treatment-induced fibrosis or necrosis, providing prognostic and therapeutic guidance.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No